CLINICAL TRIAL: NCT01716910
Title: Effect of Synbiotic on Composition of Human Gut Microbiota and Production of Short and Branched-chain Fatty Acids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Gabriella C. van Zanten, PhD student, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DK-H-4-2010-137
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Synbiotics; Healthy Humans; Composition of Gut Microbiota; Short and Branched-chain Fatty Acids
MeSH Terms: interventions — Cellobiose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator): 'Combination of Lactobacillus acidophilus NCFM and cellobiose', Sachet, 5 g/day
  Interventions: Dietary Supplement: Combination of Lactobacillus acidophilus NCFM and cellobiose
- Synbiotic (Active Comparator): 'Combination of Lactobacillus acidophilus NCFM and cellobiose', Sachet, 5 g/day + 10e9 CFU
  Interventions: Dietary Supplement: Combination of Lactobacillus acidophilus NCFM and cellobiose

INTERVENTIONS:
Dietary Supplement: Combination of Lactobacillus acidophilus NCFM and cellobiose

SUMMARY:
This is a randomized, double-blind, placebo controlled, cross-over, single centre, 14 week clinical trial on healthy volunteers. Following a two week run-in-period, subjects were randomized, and treatment with synbiotic or placebo for 21 days was given, followed by a 3-week wash-out period before the second treatment period, followed by a another wash-out period. Volunteers completed questionnaires for each period on overall health and well being, stool frequency and consistency and gastrointestinal symptoms. The subjects were asked to collect fecal samples for investigation of microbiological and microbial metabolites before and after three treatment periods. The primary objective of the study is tan increase in fecal butyrate concentration. Secondary objectives are changes in microbiota composition and short-chain fatty acids.

ELIGIBILITY:
Inclusion Criteria:healthy individuals between 18-50 years of age who had not used antibiotics three months prior to the trial

-

Exclusion Criteria:

* chronic illness
* regular intake of medication (except birth-control pills)
* post-menopausal women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
increase in fecal butyrate concentration | 12 weeks (2x 3 week intervention periods which each were followed by a 3 week wash-out period, sampling at the end of each period)

SECONDARY OUTCOMES:
changes in composition of microbiota | 12 weeks (2x 3 week intervention periods which each were followed by a 3 week wash-out period, sampling at the end of each period)
changes in short-chain fatty acids | 12 weeks (2x 3 week intervention periods which each were followed by a 3 week wash-out period, sampling at the end of each period)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella C. van Zanten, PhD student, Principal Investigator — Department of Food Science, Food Microbiology, Faculty of Science, University of Copenhagen, Denmark; Gabriella C van Zanten, PhD student, Principal Investigator — Department of Food Science, Food Microbiology, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department of Food Science, Food Microbiology, Faculty of Science, University of Copenhagen, Frederiksberg C, Denmark